CLINICAL TRIAL: NCT00191672
Title: A Phase II Randomized Trial Of Gemcitabine Plus Paclitaxel And Gemcitabine Plus Docetaxel In Patients With Metastatic Breast Cancer
Brief Title: A Trial Of Gemcitabine Plus Paclitaxel And Gemcitabine Plus Docetaxel In Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6966; B9E-US-S308
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine; Paclitaxel; Docetaxel

INTERVENTIONS:
Drug: Gemcitabine
Drug: Paclitaxel
Drug: Docetaxel

SUMMARY:
The combination of docetaxel and gemcitabine has shown significant activity in patients with metastatic breast cancer. Several studies have activity in patients of multiple lines of therapy, including patients that have been treated with prior taxane therapy. Overall responses have ranged from 30% to 79%. The major side effects of the combination chemotherapy have been neutropenia, anemia, asthenia, neuropathy, nausea, mucositis, and neutropenic fever

ELIGIBILITY:
Inclusion Criteria:

* Advanced or metastatic breast cancer
* Disease that can be measured by the physician or radiologic test.
* May have had one chemotherapy treatment for advanced or metastatic disease.
* Patients may have received any prior adjuvant chemotherapy, including taxane containing regimens, provided this treatment was completed at least 6 months prior to enrollment.
* Patients may have received prior hormone therapy or immunotherapy.

Exclusion Criteria:

* Patients with only non-measurable disease
* Cancer that has spread to the brain
* A patient who received a taxane with metastatic disease.
* Pregnancy
* Patients who received prior gemcitabine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2003-12; Study Completion 2006-11

PRIMARY OUTCOMES:
Estimate the response rate of two regimens separately.

SECONDARY OUTCOMES:
Estimate the following activities of two regimens separately:Progression-free survival;Time to progressive disease;duration of response;Overall survival, changes in performance status
Nature of toxicities experienced on each arm of the study

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CT-LILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Katy, Texas